CLINICAL TRIAL: NCT03690635
Title: Root Coverage With Connective Tissue Graft Associated With VISTA Versus Tunnel Technique in Miller Class I & II Recession Defects A Randomized Controlled Clinical Trial
Brief Title: Root Coverage With Connective Tissue Graft Associated With VISTA Versus Tunnel Technique
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mustafa Gameel Mustafa Darweesh, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio 0102051
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Root Coverage; Tunneling Technique; VISTA Technique; Sub Epithelial Connective Tissue Graft
Keywords: treatment of gingival recession; root coverage; tunneling technique; VISTA technique; sub epithelial connective tissue graft; recession treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VISTA technique (Experimental): evolution of a newer approach known as Vestibular Incision Subperiosteal Tunnel Access (VISTA) was proposed to avoid some of the potential complications occurring with other intrasulcular tunneling techniques
  Interventions: Procedure: VISTA (vestibular incision subperiosteal tunnel acess)
- tunneling technique (Active Comparator): Several modifications of tunnel technique have been described in order to preserve esthetics, avoid relapse of gingival recession and maintain papillary integrity. These modifications also attend to avoid scar formation and delayed healing related to vertical releasing incision
  Interventions: Procedure: VISTA (vestibular incision subperiosteal tunnel acess)

INTERVENTIONS:
Procedure: VISTA (vestibular incision subperiosteal tunnel acess) — A vertical incision will be made on the mucous membrane and the periosteum with a scalpel. The incision will be 8-10mm long, beginning from the mobile mucosa and reaching the apical end of the keratinized gingiva.
  A small subperiosteal elevator will be inserted through the incision and is used to free the subperiosteal tunnel flap. The flap includes the tissues of the mobile and immobile mucosa in the area of the affected teeth and about 1 mm distally and medially from them.
  Subperiosteal tunnel will be extended interproximally under each papilla as far as the embrasure space permits, without making any surface incisions through the papilla.
  Tunneling instruments will be used through the vertical incision to free the mucosa and the periosteum around the teeth affected by the gingival recession. This is continues at the base of the gingival papillae without affecting their integrity.
  Other Names: vestibular incision subperiosteal tunnel access

SUMMARY:
Several techniques were proposed in the literature to solve the problems associated with gingival recession. Root coverage was mainly indicated for esthetic concern, however, it might also be indicated for treatment of root hypersensitivity and maintaining adequate plaque control by keratinized tissue augmentation.

These proposed surgical techniques were well-documented with successful outcomes. Each technique had its own advantages, disadvantages and indications. Various factors affected the most suitable technique. These factors were either related to the dimensions of gingival recession defect, or related to the surgeon experience or to the patient himself .

Nowadays, the scope of scientific research is concerned with designing surgical techniques that are more predictable, high esthetic, less invasive and patient centered In this way, continuous modification of surgical techniques aroused to result in a more reproducible outcomes; such as the attempt to advance pedicle flaps without vertical releasing incisions, as in the modified coronally advanced flap and the modified microsurgical tunnel technique.

However, controversy still exist in the literature regarding the best technique for root coverage. Coronally advanced flap is the most commonly reported technique in research, with lack of researches on tunneling techniques.

DETAILED DESCRIPTION:
Nowadays, esthetic demands increased greatly where all seek a Hollywood smile with a white well-aligned teeth and pink healthy gingiva. Therefore, the demand on treatment of gingival recession increased. Since most gingival recession cases are generalized or involve multiple sites so, current research is focusing on how treatment of multiple recession defects can be efficient and less traumatic.

Several modifications of tunnel technique have been described in order to preserve esthetics, avoid relapse of gingival recession and maintain papillary integrity. These modifications also attend to avoid scar formation and delayed healing related to vertical releasing incision.

Although tunneling technique excluded vertical incisions with its drawbacks, tunneling was still a sensitive and a blind technique with increased trauma to sulcular epithelium which eventually resulted in unfavorable healing outcomes. So evolution of a newer approach known as Vestibular Incision Subperiosteal Tunnel Access (VISTA) was proposed to avoid some of the potential complications occurring with other intrasulcular tunneling techniques.

Moreover, a study by Cairo et al., 2009 reported increased incidence of post-operative pain and increased chair side time with tunneling in comparison to coronally advanced flap.

However, the evidence in literature is minimal on VISTA technique and there is no enough data comparing patient morbidity and root coverage outcomes between intrasulcular tunneling and vestibular tunneling except for few case reports. Therefore, this study aim to do a randomized clinical trial in order to assess the efficacy of VISTA technique in treatment of multiple gingival recession and compare it to tunneling technique.

The use of connective tissue graft seems to be a key of success in treatment of gingival recession regardless of the surgical technique used. Although there are numerous studies focusing on the effect of subepithelial connective tissue graft for the treatment of localized gingival recessions, but still more studies are needed to focus on the treatment of multiple recession defects.

Therefore, this study will monitor the effect of tunneling and VISTA techniques together with connective tissue graft on patient morbidity and root coverage outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older.
2. Periodontally and systemically healthy.
3. Presence of at least one Miller class I or II buccal gingival recession defect ≥1 and <6 mm in depth (Miller 1985)
4. Teeth to be treated: Upper and lower central and lateral incisors, canine, first and second premolars, and first molar
5. Full-mouth plaque and bleeding scores ≤ 20%, no pocket depths >3 mm, no active periodontal Disease.
6. Clinical indication and/or patient request for recession coverage.
7. Radiographic evidence of sufficient interdental bone (i.e., the distance between the crestal bone and the cementoenamel junction is not greater than two mm)
8. Gingival thickness of at least 0.5mm at a point located three mm below the free gingival margin.
9. A minimum of two mm of keratinized gingiva (thick biotype).

Exclusion Criteria:

1. Miller class III or IV recession defects.
2. Thin biotype , gingival thickness less than or equal 0.5
3. Smokers as smoking is a contraindication for any plastic periodontal surgery (Khuller, 2009).
4. Handicapped and mentally retarded patients.
5. Teeth with cervical restorations, abrasion.
6. Patients unable to undergo minor oral surgical procedures.
7. Patients with a history of drug or alcohol abuse.
8. Patients with a history of psychiatric disorder.
9. Pregnant females.
10. Uncontrolled periodontal disease or patient unwillingness to undergo needed periodontal therapy around remaining teeth.
11. Patients who have any systemic condition that may contraindicate any other surgical procedures such as bleeding disorders, uncontrolled diabetes mellitus and immune compromised patients such as HIV patients.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2020-09-10 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
post operative edema | immediately post operative
  post operative edema will be measured using visual analogue scale (VAS). Visual analogue scales (VAS) are used to measure the intensity or frequency of the symptoms and the pain. They are generally completed by patients themselves. The used scale in this study is a horizontal straight line of a fixed length (100 mm) and numbered every 10 mm ranging from "0 - no pain" to "100 - intolerable pain"

SECONDARY OUTCOMES:
Percentage of root coverage | 6 month
  Percentage of root coverage will be measured in millimeters using periodontal probe
Root Coverage Esthetic Score | 6 month
  Score (Cairo et al., 2009)

OTHER OUTCOMES:
Post-Operative Pain | immediately post operative
  post operative pain will be measured using visual analogue scale (VAS). Visual analogue scales (VAS) are used to measure the intensity or frequency of the symptoms and the pain. They are generally completed by patients themselves. The used scale in this study is a horizontal straight line of a fixed length (100 mm) and numbered every 10 mm ranging from "0 - no pain" to "100 - intolerable pain"
Gingival Thickness | 6 month
  Anesthetic Needle with a stopper (Paolantonio et al., 2002)
Gingival Recession Width (RW) | 6 month
  William's graduated Periodontal probe
Gingival Recession Depth (RD) | 6 month
  William's graduated Periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: weam battawy, PHD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
i will check with the study chair

REFERENCES:
- [Result] Gobbato L, Nart J, Bressan E, Mazzocco F, Paniz G, Lops D. Patient morbidity and root coverage outcomes after the application of a subepithelial connective tissue graft in combination with a coronally advanced flap or via a tunneling technique: a randomized controlled clinical trial. Clin Oral Investig. 2016 Nov;20(8):2191-2202. doi: 10.1007/s00784-016-1721-7. Epub 2016 Jan 27. PMID 26814715